CLINICAL TRIAL: NCT00005888
Title: Study of the Relationship Between Feeding and Late Onset Sepsis and/or Necrotizing Enterocolitis in Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/15024; BCM-H5433
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Necrotizing Enterocolitis; Sepsis
Keywords: gastrointestinal disorders; immunologic disorders and infectious disorders; low birth weight; necrotizing enterocolitis; neonatal disorders; rare disease; sepsis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis; Gastrointestinal Diseases; Immune System Diseases; Communicable Diseases; Infant, Newborn, Diseases; Rare Diseases

INTERVENTIONS:
Behavioral: Fortified Pasteurized Donor Human Milk supplement
Behavioral: Preterm Formula supplement

SUMMARY:
OBJECTIVES: I. Compare the incidence of late onset sepsis and/or necrotizing enterocolitis and duration of hospitalization in low birth weight infants fed with fortified mother's milk supplemented with either fortified pasteurized donor human milk or preterm formula, and with fortified mother's milk versus preterm formula.

II. Determine the relationship between functional antibody titers in serial milk samples and the incidence of pathogen specific late onset sepsis (e.g., Staphylococcus epidermidis, Staphylococcus aureus) in these patients.

III. Determine the long term sequelae (growth, body composition, health, and neurodevelopment) of human milk versus formula feeding in these patients.

IV. Determine the relationship between stress and milk production in the mothers of these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study in arms I and II. Patients are randomized to receive either fortified pasteurized donor human milk (arm I) or preterm formula (arm II) as a supplement to mother's milk, if needed. Patients are stratified according to gestational age (less than 26 weeks vs 27-29 weeks) and prior antenatal steroids (yes vs no). Patients are also assigned to groups receiving fortified mother's milk (arm III) and preterm formula only (arm IV).

Milk samples are obtained from the patient's mother for analyses of functional antibody against Staphylococcus epidermidis and Staphylococcus aureus; bacterial culture and sensitivity; bacterial colony count; and immunoglobulin and nutrient composition (i.e., energy, protein). Maternal blood samples to measure functional antibody are obtained every 2 weeks throughout hospitalization as long as infant is receiving own mother's milk. Cord blood is obtained at delivery.

Patients are studied at 40 week postmenstrual age, and then every 6 months for 3 years. Records of health (e.g., number of doctor, clinic, and emergency room visits; hospitalizations; and illnesses), dietary intake, and growth are collected. Urine is collected every 2 weeks to monitor infection. Neurodevelopment is assessed at 3 years using the McCarthy Scales of Infant Development.

Mothers who plan to nurse their infants after hospital discharge complete the STAI "trait" form at beginning of study. Mothers are assessed weekly for 6 weeks postpartum, and every other week thereafter as long as they are expressing milk by mechanical means only. Following a session of skin to skin contact, the number of milk expressions, the duration of each pumping, and a 24 hour milk collection is obtained. Mothers also complete the Spielberger State Trait Anxiety Inventory, STAI, Beck Depression Inventory, Norbeck Social Support questionnaire, Parental Stressor Scale, and the Neonatal Perception Inventory during each 24 hour milk collection.

ELIGIBILITY:
* Infants of less than 30 weeks gestational age
* Less than 96 hours after birth
* No HIV positive mothers who plan to nurse
* No major congenital malformations

Ages: 0 Years to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Schanler, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States